CLINICAL TRIAL: NCT06394648
Title: Investigation of Sarcopenia and Physical Fitness Levels of Geriatric Individuals Living in Nursing Homes and at Home
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Other Study IDs: E-59394181-604.01-83960
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Geriatric Individuals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Geriatric individuals living in nursing homes: Geriatric individuals living in nursing homes will be included.
- Geriatric individuals living at home: Geriatric individuals living at home will be included.

SUMMARY:
To examine the sarcopenia and physical fitness levels of geriatric individuals living in nursing homes and at home. Considering these aims, our working hypotheses are;

H1: There is a difference in sarcopenia level between geriatric individuals living in a nursing home and at home.

H2: There is a difference in dynapenia levels between geriatric individuals living in a nursing home and at home.

H3: There is a difference in physical fitness between geriatric individuals living in a nursing home and at home.

DETAILED DESCRIPTION:
Geriatric individuals living in the Nursing Home and at home will be included in the research. Within the scope of the study, anterior thigh thickness of geriatric individuals will be evaluated by ultrasonography and the presence of sarcopenia will be determined according to the Sonographic T-high Adjustment Rate (STAR) method, and the presence of dynapenia will be determined according to hand grip strength in individuals without sarcopenia. Additionally, the physical fitness of geriatric individuals in both groups will be evaluated with the Senior Fitness test. The study will be carried out with 100 geriatric individuals. As a result of the study, individuals in the groups will be compared in terms of the presence of sarcopenia and dynapenia and physical fitness.

ELIGIBILITY:
Inclusion Criteria:

* Getting a score between 24 and 30 on the Mini Mental State Exam
* Living in a nursing home for at least six months (for nursing home residents)
* Ability to stand without assistance for at least 90 seconds

Exclusion Criteria:

* Inability to communicate verbally
* Using a walking aid
* Elderly people with severe visual impairment, neurological disorders and/or congestive heart failure
* Older adults for whom exercise is not recommended

Ages: 65 Years to 85 Years | Sex: All
Age Groups: Older Adult
Study Population: Geriatric individuals
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2024-04-28 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Ultrasonography Evaluation: | Baseline
  Anterior thigh muscle thickness will be measured to evaluate sarcopenia. The obtained value will be divided by Body Mass Index (BMI). This evaluation method is referred to in the literature as the Sonographic T-high Adjustment Rate (STAR) method. Ultrasonographic measurements will be made by a physician with at least 10 years of experience in this field using linear probes.
Senior Fitness Test | Baseline
  This test evaluates the level of functional fitness at which activities of daily living can be performed safely and independently without fatigue. In daily life, physiological parameters are related to performance. Senior Fitness Test evaluates physiological parameters such as muscle strength, flexibility, aerobic endurance, balance and body composition. Senior Fitness Test consists of seven subtests and determination of body composition: Chair sit-to-stand test, weight lifting test, six-minute walk or two-minute step test, chair sit-and-reach test, back scratching test, eight-step up-to-walk test and determination of body mass index.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Principal Investigator — Atılım University; Özlem Yürük, Prof.Dr, Study Chair — Baskent University; Büşra Seçkinoğulları Korkusuz, MSc, Study Chair — Hacettepe University; Ferdi Yavuz, Assoc.Prof., Study Chair — European University of Lefke
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kara M, Kaymak B, Ata AM, Ozkal O, Kara O, Baki A, Sengul Aycicek G, Topuz S, Karahan S, Soylu AR, Cakir B, Halil M, Ozcakar L. STAR-Sonographic Thigh Adjustment Ratio: A Golden Formula for the Diagnosis of Sarcopenia. Am J Phys Med Rehabil. 2020 Oct;99(10):902-908. doi: 10.1097/PHM.0000000000001439. PMID 32941253
- [Background] Wang JC, Wu WT, Chang KV, Chen LR, Chi SY, Kara M, Ozcakar L. Ultrasound Imaging for the Diagnosis and Evaluation of Sarcopenia: An Umbrella Review. Life (Basel). 2021 Dec 22;12(1):9. doi: 10.3390/life12010009. PMID 35054402
- [Background] Kazoglu M, Yuruk ZO. Comparison of the physical fitness levels in nursing home residents and community-dwelling older adults. Arch Gerontol Geriatr. 2020 Jul-Aug;89:104106. doi: 10.1016/j.archger.2020.104106. Epub 2020 May 15. PMID 32447125